CLINICAL TRIAL: NCT07125196
Title: Incidence of Depression and Its Complications After Surgical Site Infection - ISODEP.
Acronym: ISODEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/09
Record Dates: First submitted 2025-07-07; First posted 2025-08-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Surgical Site Infections; Depression; Malnutrition
Keywords: surgical site infection; depression; malnutrition; orthopedic surgery; mood disorders; infection management; prospective study
MeSH Terms: conditions — Surgical Wound Infection; Depression; Malnutrition; Mood Disorders | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical site infection (Other): Patients treated for surgical site infection (prosthetic surgery and trauma surgery)
  Interventions: Other: Data collection and self-administered questionnaire

INTERVENTIONS:
Other: Data collection and self-administered questionnaire — Exhaustive collection of data in a health data warehouse: collection of clinical, radiological examinations (standard of care), and self-administered questionnaire: a questionnaire concerning the psychological state of the patients (questionnaire according to DSM V) and a questionnaire on nutritional status.

SUMMARY:
Surgical-site infection (SSI) in orthopedic surgery is a serious and frequent complication with many consequences on the patient's quality of life. This study aims to describe the incidence of depression and its complications like malnutrition in patients followed for surgical site infection to allow their best management and prevention

DETAILED DESCRIPTION:
We will conduct a monocentric (department orthopedic surgery, University Hospital of Bordeaux, France) prospective observational study for 5 years, involving all patients treated for surgical site infection (prosthetic surgery and trauma surgery) The data collected will concern the general condition of the patients, demographic data, information about septic condition, psychiatric disorders, or nutritional conditions, as well as the care provided. A three-year follow-up will be planned

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years old
* Patient treated in infectiology for surgical site infection after orthopedic surgery of the limbs or spine:

  * Prosthetic limb surgery
  * Spinal surgery
  * Traumatology: Osteosynthesis of peripheral limbs or spine

Exclusion Criteria:

* Patient under guardianship or curatorship,
* Pregnant, breastfeeding woman
* Person deprived of liberty by judicial or administrative decision,
* Person undergoing psychiatric treatment under duress requiring the consent of the legal representative.
* Person unable to express their consent,
* Person under legal protection,
* Patient not affiliated to a social protection scheme.
* Patient with a history of diagnosed depression, hospitalization for depressive disorders or taking mood-regulating treatments.
* An initial BMI of less than < 18.5, the existence a cancerous pathology, an ongoing inflammatory disease, a pathology responsible for chronic undernutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Depressive Episodes | Weeks 6, Month 3, Month 6 and Month 12
  Incidence of major depressive episodes as defined by the DSM V criteria, screened using the Major Depression Inventory (MDI) score. This will be assessed at baseline (M0) and at subsequent follow-up visits (Weeks 6, Month 3, Month 6 and Month 12).

SECONDARY OUTCOMES:
Socio-Demographic and Clinical Characteristics | Baseline (day 0) and 12 months (M12)
  Collection of socio-demographic data including age, sex, employment status, medical and surgical history, and smoking status at baseline and at the end of the study (M12).
Incidence of Malnutrition and Its Risk Factors | 12 months
  - Malnutrition is defined by weight loss ≥ 5% in 1 month, ≥ 10% in 6 months, or ≥ 10% compared to usual weight before illness (HAS definition); BMI < 18.5 kg/m².
Prognostic Significance of Malnutrition and Depression on Infection Treatment Efficacy and Safety | Baseline (Day 0), Week 6, Month 3, Month 6, and Month 12
  - Success of infection treatment defined by the cessation of ongoing antibiotic therapy.
Incidence of Malnutrition and Its Risk Factors | 12 months
  Monitoring current nutritional management (oral supplements, nutritional assessments conducted).
Incidence of Malnutrition and Its Risk Factors | 12 months
  - Biological criteria for malnutrition: levels of albumin, pre-albumin, folate (B9), and vitamin B12.
Incidence of Malnutrition and Its Risk Factors | 12 months
  - Assessment using the Mini Nutritional Assessment (MNA) questionnaire.
Prognostic Significance of Malnutrition and Depression on Infection Treatment Efficacy and Safety | Baseline ( Day 0), Week 6, Month 3, Month 6, and Month 12
  - Modifications in infection management due to malnutrition and depression events: treatment discontinuation, therapeutic changes.
Prognostic Significance of Malnutrition and Depression on Infection Treatment Efficacy and Safety | Baseline (Day0), Week 6, Month 3, Month 6, and Month 12
  - Quality of life scales: SF-36 (SF-36v2® Health Survey ©) and EQ-5D-5L (EuroQol Research Foundation©).
  These parameters will be assessed at baseline (Day 0) and during follow-up visits (W6, M3, M6, and M12).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin BOUYER, PROF, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France